CLINICAL TRIAL: NCT03874299
Title: The TOGETHER Project - Transplant Organ Genomics to Help Prevent Rejection in Kidney Transplant Recipients-RNA-seq Signature Validation
Brief Title: The TOGETHER Project - Kidney RNA-seq Validation
Acronym: TOGETHER
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Stegall, Principal Investigator, Mayo Clinic
Other Study IDs: 16-004433
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draws collected at 1 month, 4 month, 6 month, 9 months, 12 months and for cause.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney Transplant Receipients

SUMMARY:
The researchers are trying to develop a way to measure the risk of rejection through the validation of a blood test.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>/=18 years) renal transplant recipient.
* Patients who have given informed consent and are willing to comply with the protocol, including the use of their peripheral blood specimens and data for subsequent research.

Exclusion Criteria:

-Adult (<18 years) renal transplant recipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant recipients.
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
To validate the use of a RNA-seq based peripheral blood assay in renal transplant recipients. | 3 years
  The study will validate the ability of a peripheral blood assay to assess the risk of biopsy proven rejection.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials